CLINICAL TRIAL: NCT00079261
Title: Gem-CHOP: A Randomized Phase II Study of Gemcitabine Combined With CHOP in Untreated Aggressive Non-Hodgkin's Lymphoma
Brief Title: Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone With or Without Gemcitabine in Treating Patients With Previously Untreated Aggressive Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-20021; EORTC-20021
Record Dates: First submitted 2004-03-08; First posted 2004-03-10 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lymphoma; Small Intestine Cancer
Keywords: contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; stage III adult diffuse large cell lymphoma; stage IV adult diffuse large cell lymphoma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; adult grade III lymphomatoid granulomatosis; small intestine lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy | interventions — VAP-cyclo protocol; Cyclophosphamide; Doxorubicin; Gemcitabine; Prednisone; Vincristine

INTERVENTIONS:
Drug: CHOP regimen
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: gemcitabine hydrochloride
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, vincristine, prednisone, and gemcitabine, work in different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one chemotherapy drug may kill more cancer cells.

PURPOSE: This randomized phase II trial is studying giving combination chemotherapy together with gemcitabine to see how well it works compared to giving combination chemotherapy alone in treating patients with previously untreated aggressive stage II, stage III, or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the complete response rate (confirmed or unconfirmed) in patients with previously untreated aggressive non-Hodgkin's lymphoma treated with cyclophosphamide, doxorubicin, vincristine, and prednisone with vs without gemcitabine.

Secondary

* Compare the safety profile of these regimens in these patients.
* Compare the feasibility of these regimens, defined as the proportion of courses given as scheduled, in these patients.
* Compare freedom from treatment failure in patients treated with these regimens.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to participating center, International Prognostic Index score (0-2 vs 3-5), and histology (B cell vs T cell). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral or IV prednisone on days 1-5.
* Arm II: Patients receive CHOP chemotherapy as in arm I and gemcitabine IV over 30 minutes on days 1 and 8.

In both arms, treatment repeats every 3 weeks for 3 courses in the absence of unacceptable toxicity or progressive disease. Patients achieving partial response or complete or unconfirmed complete response receive an additional 5 courses of therapy (for a total of 8 courses).

Patients are followed every 3 months for 3 years, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 76-82 patients (38-41 per treatment arm) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive non-Hodgkin's lymphoma (NHL) of 1 of the following WHO subtypes:

  * Diffuse large B large cell lymphoma (including all clinical and morphologic variants)
  * Grade 3 follicular lymphoma
  * Extranodal T/NK cell lymphoma, nasal type
  * Enteropathy-type T cell lymphoma
  * Hepato-splenic T cell lymphoma
  * Peripheral T cell lymphoma, unspecified
  * Angioimmunoblastic lymphoma
  * Anaplastic large cell lymphoma, systemic type
* Stage II-IV disease
* At least 1 site of measurable disease (e.g., lymph node or lymph node mass)
* The following subtypes are not allowed:

  * Mantle cell lymphoma
  * Burkitt's lymphoma
  * Precursor B or T cell lymphoma
  * Primary cutaneous B or T cell lymphoma
* No CNS involvement by lymphoma

PATIENT CHARACTERISTICS:

Age

* 18 to 70

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC > 3,000/mm^3
* Neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 2.5 times normal (unless due to lymphoma)
* ALT and AST < 2.5 times normal (unless due to lymphoma)

Renal

* Creatinine < 2.0 mg/dL

Cardiovascular

* No severe cardiac disease that would preclude study participation or limit life expectancy

Pulmonary

* FEV_1 and DLCO ≥ 75% of predicted (unless due to lymphoma)
* No severe pulmonary disease that would preclude study participation or limit life expectancy

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No other prior or concurrent malignancy except basal cell skin cancer or carcinoma in situ of the cervix
* No severe neurologic or metabolic disease that would preclude study participation or limit life expectancy
* No psychological, familial, sociological, or geographical condition that would preclude study compliance and follow-up

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent monoclonal antibodies

Chemotherapy

* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy
* No concurrent radiotherapy

Surgery

* Not specified

Other

* No prior cytotoxic agents
* No prior treatment for NHL
* No other concurrent anticancer therapy
* No other concurrent investigational drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2004-01; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Complete response as assessed by Cheson criteria

SECONDARY OUTCOMES:
Toxicity as assessed by CTC 2.0
Proportion of courses given as scheduled
Freedom from treatment failure as assessed by Cheson criteria

CONTACTS AND LOCATIONS:
Overall Officials: Igor Aurer, MD, PhD, Study Chair — University Hospital Rebro
Locations (6):
- Belgium (2):
  - U.Z. Gasthuisberg, Leuven
  - Algemeen Ziekenhuis Sint-Augustinus, Wilrijk
- University Hospital Rebro, Zagreb, Croatia
- National Cancer Institute - Cairo, Cairo, Egypt
- Institut Bergonie, Bordeaux, France
- Universitair Medisch Centrum St. Radboud - Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Result] Aurer I, Eghbali H, Raemaekers J, Khaled HM, Fortpied C, Baila L, van der Maazen RW; EORTC Lymphoma Group. Gem-(R)CHOP versus (R)CHOP: a randomized phase II study of gemcitabine combined with (R)CHOP in untreated aggressive non-Hodgkin's lymphoma--EORTC lymphoma group protocol 20021 (EudraCT number 2004-004635-54). Eur J Haematol. 2011 Feb;86(2):111-6. doi: 10.1111/j.1600-0609.2010.01540.x. Epub 2010 Dec 22. PMID 20942843